CLINICAL TRIAL: NCT06500221
Title: Breathing New Life: The Impact of Incentive Spirometer Training on Rehabilitation and Health in Type 2 Diabetes With Sarcopenia
Brief Title: Incentive Spirometer Training in Type 2 Diabetes With Sarcopenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yu-Shan Hsieh (Other)
Responsible Party: Sponsor-Investigator, Yu-Shan Hsieh, Associate professor, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: N202404019
Record Dates: First submitted 2024-07-05; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes; Sarcopenia
Keywords: Type 2 diabetes; sarcopenia; incentive spirometer; lung function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sarcopenia

STUDY DESIGN:
Intervention Model Description: patients with Type 2 diabetes combined with sarcopenia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 2 diabetes combined with sarcopenia (Experimental): incentive spirometry intervention
  Interventions: Behavioral: incentive spirometry
- Type 2 diabetes combined with sarcopenia control (No Intervention): Routine care.

INTERVENTIONS:
Behavioral: incentive spirometry — The incentive spirometer is widely used in physical, speech, and respiratory therapy, as well as in preventing postoperative pulmonary infections and improving sputum clearance. Consequently, this study aims to further confirm the role and effectiveness of incentive spirometry in improving lung function, activity endurance, and long-term blood sugar and lipid indices in patients with Type 2 diabetes combined with sarcopenia.
  Arms: Type 2 diabetes combined with sarcopenia

SUMMARY:
In patients with Type 2 diabetes, the risk of developing sarcopenia is three times higher compared to individuals with normal blood sugar levels. Sarcopenia is often accompanied by reduced physical activity, immobility, slow gait, and poor endurance. More importantly, previous studies have shown that sarcopenia leads to a decrease in mobility, which in turn results in reduced cardiopulmonary function, difficulty in breathing, and subsequently even less activity. In diabetic patients, this can cause poor control of blood sugar and lipids, as well as sarcopenic obesity, creating a vicious cycle. Therefore, preventing such a cycle is a crucial issue that needs attention. The incentive spirometer is widely used in physical, speech, and respiratory therapy, as well as in preventing postoperative pulmonary infections and improving sputum clearance. Consequently, this study aims to further confirm the role and effectiveness of incentive spirometry in improving lung function, activity endurance, and long-term blood sugar and lipid indices in patients with Type 2 diabetes combined with sarcopenia.

DETAILED DESCRIPTION:
In patients with Type 2 diabetes, the risk of developing sarcopenia is three times higher compared to individuals with normal blood sugar levels. Sarcopenia is often accompanied by reduced physical activity, immobility, slow gait, and poor endurance. More importantly, previous studies have shown that sarcopenia leads to a decrease in mobility, which in turn results in reduced cardiopulmonary function, difficulty in breathing, and subsequently even less activity. In diabetic patients, this can cause poor control of blood sugar and lipids, as well as sarcopenic obesity, creating a vicious cycle. Therefore, preventing such a cycle is a crucial issue that needs attention. The incentive spirometer is widely used in physical, speech, and respiratory therapy, as well as in preventing postoperative pulmonary infections and improving sputum clearance. Consequently, this study aims to further confirm the role and effectiveness of incentive spirometry in improving lung function, activity endurance, and long-term blood sugar and lipid indices in patients with Type 2 diabetes combined with sarcopenia.

The inclusion criteria:

1. Diagnosed with Type 2 diabetes (ICD-10 diagnosis codes: E10.x or E11.x)
2. Screened with a score of 4 or above on the screening self-administered sarcopenia (SARC-F) questionnaire.
3. Aged between 20-90 years old and able to communicate in Mandarin or Taiwanese

The exclusion criteria:

1. Patients with a functional status grade of ≥5 on the Modified Rankin Scale (MRS), indicating severe disability or bedridden condition.
2. Patients suffering from dementia, such as Alzheimer's disease, Parkinson's disease, etc.
3. Patients with acute psychiatric symptoms unable to communicate.
4. Currently diagnosed with chronic obstructive pulmonary disease (COPD) or any other respiratory system diseases.
5. Moderate or severe heart disease (New York Heart Association functional classification Class III or IV).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 diabetes (ICD-10 diagnosis codes: E10.x or E11.x)
* Screened with a score of 4 or above on the SARC-F questionnaire.
* Aged between 20-90 years old and able to communicate in Mandarin or Taiwanese

Exclusion Criteria:

* Patients with a functional status grade of ≥5 on the Modified Rankin Scale (MRS), indicating severe disability or bedridden condition.
* Patients suffering from dementia, such as Alzheimer's disease, Parkinson's disease, etc.
* Patients with acute psychiatric symptoms unable to communicate.
* Currently diagnosed with chronic obstructive pulmonary disease (COPD) or any other respiratory system diseases.
* Moderate or severe heart disease (New York Heart Association functional classification Class III or IV).

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Lung function: FVC | 3 months
  Forced Vital Capacity (FVC)
Lung function:FEV1 | 3 months
  Forced Expiratory Volume in the First Second (FEV1)
Lung function: FEV1/FVC ratio | 3 months
  FEV1/FVC ratio

SECONDARY OUTCOMES:
Long-term Metabolic Indicators: HbA1c | 3 months
  Glycated Hemoglobin (HbA1c)
Long-term Metabolic Indicators: TG | 3 months
  Serum Triglycerides (TG)
Long-term Metabolic Indicators: LDL | 3 months
  Serum Low-Density Lipoprotein (LDL)
Long-term Metabolic Indicators: HDL | 3 months
  Serum High-Density Lipoprotein (HDL)
Long-term Metabolic Indicators: TC | 3 months
  Serum Total Cholesterol (TC)

IPD SHARING:
Plan to Share IPD: No